CLINICAL TRIAL: NCT06173908
Title: Department of Burn Surgery, The First Affiliated Hospital of Sun Yat-sen University
Brief Title: Autologous Epidermal Cell Treat for Nonhealing Postoperative Wound
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Zhu Jiayuan, Professor, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SYSU-FAH-2019286
Record Dates: First submitted 2023-12-07; First posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Healing Wound

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cell treatment (Experimental): Autologous epidermal basal cells were used to treat postoperative nonhealing wounds
  Interventions: Procedure: cell treatment
- control treatment (Sham Comparator): Conventional method were used to treat postoperative nonhealing wounds
  Interventions: Procedure: control treatment

INTERVENTIONS:
Procedure: cell treatment — Autologous epidermal basal cells were used to repair nonhealing postoperative wound
  Arms: cell treatment
Procedure: control treatment — anyother treatments except autologous epidermal basal cells were used to repair nonhealing postoperative wound
  Arms: control treatment

SUMMARY:
Postoperative incision healing (Postoperative incision non - ranging) occurred in the surgical incision more than 2 weeks after the operation is still not healing wounds.

At present, direct suture, autologous skin graft transplantation, conventional dressing change and negative pressure wound therapy are still the first-line treatment options for postoperative wound nonunion. However, the wound healing time is long and the wound healing rate is low. Autologous epidermal basal cell suspension is derived from the basal layer of the epidermis and contains 1-10% epidermal stem cells. Therefore, we plan to carry out a multi-center, prospective randomized controlled clinical trial, aiming to verify whether this technique can promote wound healing.

DETAILED DESCRIPTION:
Postoperative incision healing (Postoperative incision non - ranging) occurred in the surgical incision more than 2 weeks after the operation is still not healing wounds, show the incision infection, effusion, hemorrhage, empyema, skin lesions and skin defect. It has a high morbidity and the treatment cycle is long, the social and economic burden is heavy.

At present, direct suture, autologous skin graft transplantation, conventional dressing change and negative pressure wound therapy are still the first-line treatment options for postoperative wound nonunion. However, the wound healing time is long and the wound healing rate is low. Therefore, how to improve the wound healing rate is an urgent problem to be solved. The present study indicated that the disturbance of wound microenvironment was the main reason for the wound healing. Autologous epidermal basal cell suspension is derived from the basal layer of the epidermis and contains 1-10% epidermal stem cells. Therefore, we plan to carry out a multi-center, prospective randomized controlled clinical trial, aiming to verify whether this technique can promote wound healing.

ELIGIBILITY:
Inclusion Criteria:

* (1) the age of the subject on the day of signing the informed consent is 18 years old or above;

  (2) the diagnosis was non-union of incision, and the diagnosis criteria of non-union of incision were as follows: non-union of incision > for 2 weeks after various surgeries;

  (3) patients with stable vital signs, who are proved to be tolerable to surgery by routine examination;

  (4) the patient is in good mental state, can follow the doctor's advice and return to the hospital regularly;

  (5) understand and willing to participate in this clinical trial and provide the signed informed consent

Exclusion Criteria:

* (1) local wound complicated with malignant tumor;

  (2) during the screening period, patients showed immunosuppression due to potential diseases, long-term immunosuppressive therapy or the use of large doses of glucocorticoid (i.e.

  (3) patients with mental diseases;

  (4) patients with serious uncontrolled diseases or acute systemic infections and other serious visceral diseases such as heart, lung and brain diseases;

  (5) if the researcher considers the inclusion inappropriate;

  (6) the patients were pregnant women, fertile women who did not take appropriate contraceptive measures, lactating women during the screening period or women who planned to become pregnant within 1 month after the end of the study;

  (7) the patient participated in this study at any time in the past and the patient is participating in other clinical trials.

Max Age: 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
healing rate | postoperative day 7, 14, 21, 28
  wound healing rate

SECONDARY OUTCOMES:
healing time | when the wound was complete healed，through study completion, an average of 1 or 2 weeks
  wound healing time
recurrence rate | postoperative month 3
  recurrence rate
Wound reduction rate | postoperative day 7, 14, 21, 28
  Wound reduction rate

CONTACTS AND LOCATIONS:
Overall Officials: Jiayuan Zhu, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- Jiayuan Zhu, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No